CLINICAL TRIAL: NCT04175782
Title: Comparison of Enhanced Recovery Protocol With Conventional Care in Patients Undergoing Urogynecologic Surgery
Brief Title: Enhanced Recovery Protocol in Urogynecologic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Gulseren Yilmaz, Principal Investigator, M.D., Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gulseren4
Record Dates: First submitted 2019-11-20; First posted 2019-11-25 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Urinary Incontinence; Cystocele; Rectocele; Pelvic Organ Prolapse
MeSH Terms: conditions — Urinary Incontinence; Cystocele; Rectocele; Pelvic Organ Prolapse | interventions — Enhanced Recovery After Surgery; Clinical Protocols

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS group (Experimental): A standardized ERAS protocol is applied to the ERAS group based on the latest guidelines. Smoking and alcohol consumption is stopped 4 weeks before the surgery. Preoperative anemia is corrected with intravenous iron supplementation. Prolonged fasting, bowel preparation, and premedication are avoided in this group. Clear fluids are allowed up to 2 h and solids rich in carbohydrate up to 6 h hours prior to induction of anesthesia. Warmed up intravenous fluids are administered to maintain normothermia intraoperatively. This group of subjects receives general anesthesia. Volume and salt overload and drain usage are avoided to the utmost. Intravenous paracetamol is administered for postoperative analgesia before the completion of the surgical procedure. Nasogastric tube placement is avoided and catheters are removed as soon as possible. Nonopioid oral analgesics and NSAIDs are utilized for postoperative pain medication.
  Interventions: Procedure: Enhanced recovery after surgery (ERAS) protocol
- Control (No Intervention): This group will receive conventional pre-and postoperative care.

INTERVENTIONS:
Procedure: Enhanced recovery after surgery (ERAS) protocol — Preoperative:
  Counseling before hospital admission Fluid, and carbohydrate loading Avoiding prolongation of the fasting period Avoiding bowel preparation or its application only in selective cases Application of antibiotic prophylaxis Application of thromboprophylaxis Avoiding premedication
  Intraoperative:
  Use of short-acting anesthetic agents Refraining from using drains Refraining from salt, and water overload Maintenance of normothermia (heating the body, and use of warmed up intravenous fluids)
  Postoperative:
  Refraining from the use of nasogastric tube Prevention of nausea, and vomiting Refraining from salt, and water overload Earlier removal of catheters Initiation of oral intake at an early period Use of nonopioid oral analgesics/NSAIDs Early mobilization Adherence to the protocol, and auditing results
  Arms: ERAS group

SUMMARY:
Enhanced recovery after surgery (ERAS) has been shown to improve postoperative outcomes in a variety of surgical conditions. However, data regarding its role in urogynecologic surgery is limited. This study aimed to investigate the role of the ERAS protocol on postoperative outcomes in patients undergoing urogynecologic surgery.

DETAILED DESCRIPTION:
Enhanced recovery after surgery (ERAS) or in other words "fast-track" protocol roughly purposes to improve patient satisfaction, reduce complications and shorten the hospital stay. Chronic diseases, nutrition, and any volume depletion are corrected prior to surgery and less invasive surgical techniques are utilized to this end The impact of ERAS protocols in decreasing length of stay (LOS), reducing postoperative pain, improving early ambulation and decreasing the rate of potentially serious medical complications have been studied in patients undergoing colorectal, urologic, gastric and pancreatic surgery previously. However, data regarding the role of ERAS protocol in improving postoperative outcomes and postoperative compliance in patients undergoing urogynecological surgery is limited.

The present study purposes to clarify the role of the ERAS protocol on postoperative outcomes in patients undergoing urogynecologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age must be > 18 years
* Must be scheduled for urogynecologic surgery

Exclusion Criteria:

* Emergency surgery
* Presence of preoperative sepsis
* Presence of advanced liver or kidney disease

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Time to ambulation | Up to 1 week
  Hours

CONTACTS AND LOCATIONS:
Overall Officials: Gulseren Yilmaz, MD, Principal Investigator — Kanuni Sultan Suleyman Hospital
Locations (1):
- Kanuni Sultan Suleyman Training and Research Hospital, Istanbul, Please Enter the State Or Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No